CLINICAL TRIAL: NCT00244920
Title: An Open Label Randomized Phase 2 Study To Evaluate The Activity, Tolerability, And Toxicity Of Combined Neoadjuvant Anti-angiogenesis and Androgen Ablation Therapy in Men Undergoing Radical Prostatectomy
Brief Title: Hormone Therapy With or Without Squalamine Lactate in Treating Patients Who Are Undergoing a Radical Prostatectomy for Locally Advanced Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew drug.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000446087; OHSU-MSI-1256F-204; OHSU-IRB-357
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Leuprolide; squalamine lactate; Chemotherapy, Adjuvant; Androgen Antagonists; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bicalutamide
Drug: leuprolide acetate
Drug: squalamine lactate
Procedure: adjuvant therapy
Procedure: antiandrogen therapy
Procedure: antiangiogenesis therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: releasing hormone agonist therapy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as leuprolide and bicalutamide, may stop the adrenal glands from making androgens. Squalamine lactate may stop the growth of prostate cancer by blocking blood flow to the tumor. Giving hormone therapy together with squalamine lactate before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase II trial is studying how well giving hormone therapy together with squalamine lactate works compared to hormone therapy alone in treating patients who are undergoing a radical prostatectomy for locally advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of neoadjuvant androgen-ablation therapy with vs without squalamine lactate on induced tumor regression and grade migration in patients with locally advanced high-risk adenocarcinoma of the prostate undergoing a radical prostatectomy.
* Compare the duration of clinical disease-free survival of patients treated with these regimens.
* Determine the applicability of prostate-specific antigen (PSA) serology as an endpoint determinant in patients treated with these regimens.
* Compare the feasibility and potential safety effects on wound healing and recovery in patients treated with these regimens before and after a radical prostatectomy.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive leuprolide intramuscularly once a month for 3 months and oral bicalutamide once a day for 2 weeks.
* Arm II: Patients receive leuprolide and bicalutamide as in arm I plus squalamine lactate IV over 4 hours once weekly for 6 weeks.

Seven weeks after beginning treatment, patients in both arms undergo standard radical prostatectomy. Patients then continue to receive leuprolide and bicalutamide with or without squalamine lactate for up to 6 additional weeks.

After completion of study treatment, patients are followed periodically for at least 3 years.

PROJECTED ACCRUAL: A total of 132 patients (66 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Locally advanced disease

    * No metastatic disease
* High-risk characteristics, meeting ≥ 1 of the following criteria:

  * Large, hard tumor on digital exam
  * Aggressive-appearing cancer cells on biopsy
* Prostate-specific antigen > 10 ng/mL

PATIENT CHARACTERISTICS:

Performance status

* 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 11.0 g/dL

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* SGOT and SGPT < 2 times ULN
* PT and PTT normal

Renal

* Creatinine < 1.8 g/dL

Cardiovascular

* No history of ventricular arrhythmia or dysfunction
* No congestive heart failure
* No symptomatic coronary artery disease
* No prior myocardial infarction
* No history of thromboembolic disease (e.g., deep vein thrombosis or stroke) within the past 12 months
* No other significant cardiovascular disease

Pulmonary

* No pulmonary embolism within the past 12 months
* No exercise-limiting respiratory disease

Other

* Fertile patients must use effective barrier method contraception
* No sexual intercourse for 6 weeks after surgery
* No uncontrolled diabetes
* No serious acute infection
* No other malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior squalamine lactate

Chemotherapy

* No prior chemotherapy for prostate cancer
* No concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent systemic corticosteroids

Radiotherapy

* No prior radiotherapy for prostate cancer
* No concurrent radiotherapy

Surgery

* No prior surgery for prostate cancer
* No other concurrent surgery

Other

* At least 6 weeks since prior and no concurrent use of over-the-counter or herbal drugs that have estrogenic activity
* No participation in another investigational study within the past 3 months
* No concurrent participation in another investigational study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Tumor response in terms of tumor volume as measured by transrectal ultrasound before and after neoadjuvant treatment
Tumor response in terms of conventional histopathology as measured by prostatectomy specimens and Gleason scores in comparison to pre-treatment biopsies
Tumor response in terms of molecular markers as measured by changes in VEGF, VEGF-flt-1, and integrin Alpha6Beta4, AlphaVBeta3, and AlphaVBeta5 expression in pre-treatment biopsy and post-treatment prostatectomy specimens

SECONDARY OUTCOMES:
Safety, feasibility, and tolerability as measured by CTCAE v3.0
Prostate-specific antigen (PSA) serology as measured by PSA value during and after completion of study treatment
Survival for up to 3 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Sokoloff, MD, FACS, Study Chair — OHSU Knight Cancer Institute